CLINICAL TRIAL: NCT00685386
Title: A Randomized, Controlled, Double-blind Trial of CO2 Versus Air Insufflation During Endoscopic Retrograde Cholangiopancreatography
Brief Title: A Randomized Controlled Trial (RCT) of Carbon Dioxide Versus Air Insufflation During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Olympic Medical (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Evan S. Dellon, MD, University of North Carolina-Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 07-1404
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2011-04

CONDITIONS: Cholestasis
Keywords: endoscopic retrograde cholangiopancreatography; carbon dioxide; randomized controlled clinical trial
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental)
  Interventions: Other: CO2 insufflation
- II (Placebo Comparator): Room air will be used for insufflation as the placebo comparator arm.
  Interventions: Other: Room air insufflation

INTERVENTIONS:
Other: CO2 insufflation — The bowel lumen will be insufflated with CO2 during the endoscopy (as compared to room air).
  Other Names: Olympus XUCR manufacured by Olympus Medical.
  Arms: I
Other: Room air insufflation — During the ERCP, room air will be insufflated (current standard clinical practice) as a placebo comparator.
  Arms: II

SUMMARY:
The purpose of this study it to conduct a randomized, controlled, double-blinded trial of carbon dioxide (CO2) versus air insufflation during endoscopic retrograde cholangiopancreatography (ERCP).

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* referred for ERCP for any indication at UNC Hospitals

Exclusion Criteria:

* age < 18 years
* COPD requiring oxygen or with known CO2 retention
* any medical condition with known CO2 retention
* medical instability making the procedure unsafe
* absolute requirement for same-day second endoscopy
* ERCP performed in the OR or under GA
* inability to read or understand English
* use of chronic opiates for pain
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Abdominal pain (VAS). | pre-procedure and up to 24 hours post-procedure.

SECONDARY OUTCOMES:
The extent of CO2 retention. | Intra-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Evan S. Dellon, MD MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Dellon ES, Velayudham A, Clarke BW, Isaacs KL, Gangarosa LM, Galanko JA, Grimm IS. A randomized, controlled, double-blind trial of air insufflation versus carbon dioxide insufflation during ERCP. Gastrointest Endosc. 2010 Jul;72(1):68-77. doi: 10.1016/j.gie.2010.01.041. Epub 2010 May 20. PMID 20493485